CLINICAL TRIAL: NCT05837091
Title: Impact of Low Sodium Oxybate on Total Sleep Time in Patients With Idiopathic Hypersomnia
Brief Title: Low Sodium Oxybate in Patients With Idiopathic Hypersomnia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chad M. Ruoff, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-006906
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — Calcium; Magnesium; Potassium; Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Low Soduim Oxybate for Idiopathic Hypersomnia (Experimental): Subjects prescribed with low sodium oxybate for idopathic hypersomnia will have a 24-hour polysomnography, wear an Axivity wristband and Nextsense EEG earbuds to evaluate total sleep time.
  Interventions: Drug: Low Sodium Oxybate; Diagnostic Test: 24-hour polysomnography; Device: Nextsense EEG earbuds; Device: Axivity device

INTERVENTIONS:
Drug: Low Sodium Oxybate — Titrated according to standard of care and continued on stable dose for 3 months
  Other Names: Xywav; Calcium, Magnesium, Potassium, and Sodium Oxybates
Diagnostic Test: 24-hour polysomnography — Performed in a sleep study lab, recording of body functions including brain activity, eye movements, muscle activity, heart rhythm and blood oxygen levels while asleep and awake for a 24-hour period
Device: Nextsense EEG earbuds — Ear buds used to record sleep staging worn for a 24-hours period
Device: Axivity device — Wristband that records activity level worn for approximately one month to track sleep and steps/activity.

SUMMARY:
Low sodium oxybate has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of idiopathic hypersomnia. In this study, the researchers want to learn how low sodium oxybate impacts ability of people diagnosed with idiopathic hypersomnia to sleep for long periods of time. In addition, this study will use novel tools to determine when an individual is awake or asleep.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of IH, according to ICSD-3 criteria (does not require MSLT)
2. Subjects aged 18 - 65 years
3. BMI between 18 and 35 kg/m2
4. Self-reported sleep duration ≥ 9 hours most days including daytime naps/sleep based upon at least 10/14 days of completed sleep diary entries
5. Epworth Sleepiness Scale (ESS) ≥ 10 (required at pre-screening visit only)
6. Recommended LSO by a clinical sleep specialist as part of routine medical care. The clinical sleep specialist will be responsible for titrating LSO according to standard of care.
7. Subject must be willing to postpone LSO therapy until all baseline assessments completed
8. If treated with wake promoting agents, traditional stimulants and/or antidepressant(s), a stable dose and regimen will be required for at least 2 months before study entry and throughout the main study
9. Have used a medically acceptable method of contraception for at least 2 full menstrual cycles before participating in this study and consent to use a medically acceptable method of contraception from the first dose of study drug, throughout the entire study period, and for 30 days after the last dose of study drug.

Exclusion Criteria:

1. Succinic semialdehyde dehydrogenase deficiency, porphyria
2. Other central nervous system diseases: neurodegenerative diseases, , seizure disorders or history of head trauma associated with loss of consciousness
3. Lifetime history of suicide attempt or suicidal ideation in the past six months, including answer to question #9 on PHQ-9 ≥1; PHQ-9 total score > 10; prior history of psychotic episodes; active major depressive disorder
4. Change to psychiatric medication(s)/stimulant(s) within last 3 months
5. History of chronic alcohol or drug abuse within the prior 12 months
6. Malignant neoplastic disease requiring therapy within the prior 12 months
7. Heart failure, severe hypertension or other cardiovascular disease compromising the patient's well-being or ability to participate in this study
8. Renal or hepatic impairment
9. Compromised respiratory function (e.g., history of COPD, pulmonary hypertension, and/or poorly controlled asthma)
10. Diagnosis of sleep-related breathing disorders (AHI ≥ 15 events/h using 4 % AHI) or high suspicion for sleep disordered breathing
11. Any sleep apnea treatment (e.g., Positive Airway Pressure (PAP) therapy, oral appliance therapy, etc.)
12. No regular sleep at night: shift work or other continuous, non-disease-related life conditions
13. Participation in another study of an investigational drug within the 28 days prior to Screening visit or currently
14. Pregnant and/or breast-feeding
15. Ear jewelry and/or piercings that subject not willing to/unable to remove
16. Use of device/implant that may interfere with the study devices/procedures (e.g., vagal nerve stimulator)
17. Smoke and/or use of smokeless tobacco products
18. Subjects who, in the opinion of the investigator(s), may not be suitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Total Sleep Time | Baseline, 3 months
  Measured by the 24-hour polysomnography reported as total minutes a participant is deemed sleeping.

SECONDARY OUTCOMES:
Change in total sleep time as measured by Nextsense EEG earbuds | Baseline, 3 months
  Measured by the Nextsense EEG earbuds reported as total minutes a participant is deemed sleeping.
Change in total sleep time as measured by Axivity device | Baseline, 3 months
  Measured by the Axivity device reported as total minutes a participant is deemed sleeping.
Change in total sleep time as measured by patient sleep diary | Baseline, 3 months
  Measured by patient sleep diary entries as total minutes a participant reported sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Ruoff, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Stanford University, Redwood City, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20548952